CLINICAL TRIAL: NCT04123990
Title: Study of the Prevalence of Iron Deficiency in Patients With Chronic Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: VIFORFRANCE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CARENFER MICI
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Intestinal Disease
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBD (Experimental)
  Interventions: Diagnostic Test: Iron status testing

INTERVENTIONS:
Diagnostic Test: Iron status testing — Iron status testing

SUMMARY:
Despite its known prevalence in IBD, a recent study conducted with Prof. Cacoub (unpublished) on the national health insurance database showed that iron deficiency was an under-diagnosed and under-treated co-morbidity. In chronic diseases including IBD, Transferrin Saturation Factor is only performed in approximately 10% of cases, whereas it is recommended in inflammatory situations including IBD patients (HAS 2011).

The objective of this study is therefore to obtain updated French data on the prevalence of iron deficiency in patients with IBD by applying the recommendations of ECCO and French Health High Authority (determination of ferritinemia and Transferrin Saturation Factor)

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old
* Patient present at the hospital on the day of the study
* Diagnosis of IBD on international criteria
* Patient giving written consent

Exclusion Criteria:

* Protected patient: major under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision;
* pregnant, lactating or parturient woman;
* Patient hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2019-11-02 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Ferritinemia according to inflammatory status | One day
  Ferritinemia will be assessed from blood sample (iron status)

IPD SHARING:
Plan to Share IPD: No